CLINICAL TRIAL: NCT00587067
Title: A Phase II Study of Continuous Hepatic Arterial Infusion With Floxuridine (FUDR) and Dexamethasone (DEX) in Patients With Unresectable Primary Hepatic Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-120; NCT00310102 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Hepatic Cancer
Keywords: FUDR; FLOXORUIDINE; DEXAMETHASONE; Hepatic; Cancer; 02-120
MeSH Terms: conditions — Liver Neoplasms; Neoplasms | interventions — Floxuridine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: FLOXURIDINE

INTERVENTIONS:
Drug: FLOXURIDINE — [0.16* mg/kg/day X 30 ml] / pump flow rate
  * If the patient is >25% above ideal body weight, the dose of FUDR will be calculated from an average of the patients actual and ideal body weights. For example, for a patient who is 5ft. 10 inches and weighs 100kg: Ideal Body Weight (kg) = 50 + (2.3 X height in inches over 5 feet) = 50 + (2.3 X 10) = 73 Weight Used for dose calculation = (100 + 73)/2 = 86.5 Therefore, FUDR Dose will be = (0.16 X 86.5 X 30)/Flow Rate If no dose modification due to toxicity is required, the dosages given above (adjusted for changes in weight and pump flow rate) will be repeated on Day 1 of Week 1 of Cycle 2 and all subsequent cycles.
  Other Names: FUDR

SUMMARY:
This phase II study aims to evaluate regional chemotherapy in patients with unresectable primary hepatic malignancy. Specifically, eligible patients with hepatocellular carcinoma and peripheral cholangiocarcinoma, considered unresectable after review by the Hepatobiliary Surgery service, will undergo hepatic artery pump placement and continuous infusion of FUDR. The protocol includes radiological and biological correlative studies.

DETAILED DESCRIPTION:
This phase II study aims to evaluate regional chemotherapy in patients with unresectable primary hepatic malignancy. Specifically, eligible patients with hepatocellular carcinoma and peripheral cholangiocarcinoma, considered unresectable after review by the Hepatobiliary Surgery service, will undergo hepatic artery pump placement and continuous infusion of FUDR. The protocol includes radiological and biological correlative studies.

The primary objectives of the study are 1.) to assess the efficacy of continuous hepatic arterial infusion (HAI) of FUDR and dexamethasone (DEX) in patients with unresectable hepatocellular carcinoma (HCC) and intrahepatic cholangiocarcinoma (ICC) and 2.)to assess patient tolerability of this therapy stratified by degree of underlying hepatic parenchymal disease, as determined on liver biopsy. Secondary objectives are 1.) to use dynamic MRI to evaluate changes in tumor perfusion during treatment and to correlate these findings with radiographic tumor response and 2.) to investigate molecular genetic changes associated with these tumors using comparative genomic hybridization and cDNA array from tumor and liver biopsy specimens obtained at the time of operation. All patients enrolled in the study will begin HAI FUDR at 0.16 mg/kg/day. An initial cohort of 12 patients will be enrolled and treated. Dose limiting toxicity (DLT) related to FUDR is defined by changes in liver function blood tests that are unrelated to disease progression or mechanical biliary obstruction. Modifications in the FUDR dose may be required. A patient will be considered intolerant of therapy if treatment must be stopped due to DLT at least once during the first 3 months. Treatment will continue as long as there is at least stable disease and acceptable toxicity.

If, in the initial cohort, 4 or more patients (> 30%) are intolerant of therapy or if there are not at least 2 responders, then the study will be terminated. Otherwise, accrual will continue to a maximum of 35 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a liver mass that is radiographically consistent with HCC and a serum alpha fetoprotein (AFP) > 500 ng/dl do not require biopsy confirmation of the diagnosis.
* Patients with HCC or ICC undergoing exploration for a possible curative resection but found to have unresectable disease confined to the liver will be eligible, provided that no intraoperative findings would exclude them and prior informed consent has been obtained (see below).
* There must be <70% liver involvement by cancer, and the disease must be considered unresectable.
* Patients who have failed ablative therapy will be eligible.
* Patients must have a KPS > 60% and be considered candidates for general anesthesia and hepatic artery pump placement.
* Patients with chronic hepatitis and/or cirrhosis are eligible
* Serum albumin must be >2.5 g/dl and total serum bilirubin must be <1.8 mg/dl based on preoperative laboratory values within 14 days of registration.
* WBC must be >3500 cells/mm3 and platelet count must be >100,000/mm3 based on preoperative laboratory values within 14 days of registration.
* The international normalized ratio (INR) must be less than 1.5 in patients not on coumadin therapy, based on preoperative laboratory values within 14 days of registration.
* Age >_ 18 years.
* Female patients cannot be pregnant or lactating.
* Patients must be able to understand and sign informed consent.

Exclusion Criteria:

* Patients who have received prior treatment with FUDR
* Patients who have had prior external beam radiation therapy to the liver.
* Patients who have a diagnosis of sclerosing cholangitis.
* Patients who have a diagnosis of Gilbert's disease.
* Patients who have clinical ascites
* Patients with hepatic encephalopathy
* Patients who have radiographic evidence of esophageal varices or history of variceal hemorrhage.
* Patients with occlusion of the main portal vein nor of the right and left portal branches Patients that have concurrent malignancies (except localized basal cell or squamous cell skin cancers). Patient with active infection. Female patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-06; Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 6/24/2003, Protocol Closed to Accrual 7/24/2007, Primary Completion Date 5/19/2016, Recruitment location is the medical clinic
Groups:
- Floxuridine + Dexamethasone: FLOXURIDINE: [0.16* mg/kg/day X 30 ml] / pump flow rate
  * If the patient is >25% above ideal body weight, the dose of FUDR will be calculated from an average of the patients actual and ideal body weights. For example, for a patient who is 5ft. 10 inches and weighs 100kg: Ideal Body Weight (kg) = 50 + (2.3 X height in inches over 5 feet) = 50 + (2.3 X 10) = 73 Weight Used for dose calculation = (100 + 73)/2 = 86.5 Therefore, FUDR Dose will be = (0.16 X 86.5 X 30)/Flow Rate If no dose modification due to toxicity is required, the dosages given above (adjusted for changes in weight and pump flow rate) will be repeated on Day 1 of Week 1 of Cycle 2 and all subsequent cycles.
Period: Overall Study
Arm/Group | Floxuridine + Dexamethasone
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Floxuridine + Dexamethasone
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 56.5 [30 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: To assess the efficacy of continuous arterial infusion (HAI) of FUDR (Floxuridine) and dexamethasone (DEX) in patients with unresectable hepatocellular carcinoma (HCC) and intrahepatic cholangiocarcinoma (ICC).
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Floxuridine + Dexamethasone: Patients with hepatocellular carcinoma and peripheral cholangiocarcinoma, considered unresectable after review by the Hepatobiliary Surgery service will undergo hepatic artery pump placement and continuous infusion of Floxuridine.
Arm/Group | Floxuridine + Dexamethasone
Number analyzed (Participants) | 34
Participants
  Partial Response | 16
  Stable Disease | 14
  Progression of Disease | 4

2. Primary Outcome: Number of Patients With Treatment Related Toxicity
Description: Toxicity evaluated and graded according to the National Cancer Institute, CTCAE v4.0
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Floxuridine + Dexamethasone
Number analyzed (Participants) | 34
participants | 34

3. Secondary Outcome: Disease Progression
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Floxuridine + Dexamethasone
Number analyzed (Participants) | 34
Participants
  PD in the liver, alone | 18
  PD in the liver and an extrahepatic location | 3
  PD initially at an extrahepatic site only | 12
  No PD | 1

4. Secondary Outcome: Median Survival
Description: Median Survival from Initiation of Hepatic Arterial Infusion
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Floxuridine + Dexamethasone
Number analyzed (Participants) | 34
months | 29.3 [26.6 to 31.9]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Floxuridine + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 33/34
Serious Adverse Events (participants affected / at risk) | 5/34
Other Adverse Events (participants affected / at risk) | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Floxuridine + Dexamethasone (N=34)
Bilirubin Increased (Investigations) | 2
GI, other (Gastrointestinal disorders) | 1
Hepatic, other (Hepatobiliary disorders) | 1
Melena (Gastrointestinal disorders) | 1
Pain, other (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Floxuridine + Dexamethasone (N=34)
Increased bilirubin (Investigations) | 3
Headache/Migraine (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Wound infection (Infections and infestations) | 3
Delerium (Psychiatric disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes